CLINICAL TRIAL: NCT07113743
Title: Part B- Phase I/II, Non-Randomized, Single Site Study, Open-label Study of G1XCGD (Lentiviral Vector Transduced CD34+ Cells) in Patients With X-Linked Chronic Granulomatous Disease
Brief Title: Part B- G1X-CGD (Lentiviral Vector Transduced CD34+ Cells) in Patients With X-Linked Chronic Granulomatous Disease
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000186; 000186-I
Record Dates: First submitted 2025-08-08; First posted 2025-08-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-26

CONDITIONS: Chronic Granulomatous Disease (CGD)
Keywords: Gene Therapy; UCLA; CGD
MeSH Terms: conditions — Granulomatous Disease, Chronic | interventions — Busulfan; tocilizumab; eltrombopag; Sirolimus; Genes

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- X-linked CGD (Experimental): Non-randomized single arm
  Interventions: Drug: Busulfan; Drug: Tocilizumab; Drug: Eltrombopag; Drug: Sirolimus; Other: pCCLChimGp91lentiviral vector containing the human gp91 phox (CYBB) gene

INTERVENTIONS:
Drug: Busulfan — Conditioning drug
Drug: Tocilizumab — Monoclonal Antibody
Drug: Eltrombopag — Thrombopoietin Receptor Agonist
Drug: Sirolimus — Post transplant immunosuppressant drug
Other: pCCLChimGp91lentiviral vector containing the human gp91 phox (CYBB) gene — Intervention Infusion on Day 0

SUMMARY:
Background:

X-Linked Chronic Granulomatous Disease (X-CGD) is caused by a gene mutation that makes the immune system to not work properly. Researchers want to see if a lentiviral gene transfer treatment will have the ability to make the patient s immune system more normal, in particular reduce the risk of CGD related infections. The gene transfer takes a person s own stem cells, cultures them to put the normal gene in, then gives the cells back to the person.

Objective:

To test a gene transfer treatment for X-CGD.

Eligibility:

Participants aged 3-60 with X-CGD

Design:

Participants will be screened under protocol 05-I-0123. They will undergo:

Medical history

Physical exam

Heart tests

Imaging tests, as needed

Blood tests

Lung function tests, as needed

Dental and audiology exams, if needed

Quality of life questionnaire

Bone marrow aspiration. A needle will be inserted into the hip bone or breastbone to collect bone marrow.

Some screening tests will be repeated during the study.

Participants will have an apheresis procedure under protocol 94-I-0073. Stem cells will be collected.

Participants will get a series of drugs to prepare them for the gene transfer.

Participants will stay at the NIH Clinical Center for a little over a month. They will get a central line. It is a large intravenous (IV) catheter that is placed into a vein of the neck, chest, or arm. They will get chemotherapy and their corrected stem cells through their IV line.

Participants will have 12 follow-up outpatient visits in the 2 years after their gene transfer, as well as visits with their local doctor. Then they will enroll in another study for long-term follow-up visits that will last for 13 years.

DETAILED DESCRIPTION:
Study Description:

This is a Phase I/II, non-Randomized, Single site study, open-label study of a single infusion of autologous CD34+ cells transduced ex vivo with pCCLChimGp91/VSVg lentiviral vector in 10 patients with X-Linked CGD.

Objectives:

Primary Objective:

To evaluate the safety, efficacy and stability by biochemical and functional reconstitution in progeny of engrafted cells at 12 months Secondary Objectives:

Endpoints:

* Clinical efficacy and longitudinal evaluation of clinical effect in terms of augmented immunity against bacterial and fungal infection
* Determine the number of days of antibiotic usage before compared to after gene therapy
* Transduction efficiency of CD34+ hematopoietic cells from XCGD patients by ex vivo lentivirus-mediated gene transfer
* Evaluation of engraftment kinetics and stability

Primary Endpoint:

1. The primary safety objective of this procedure will be assessed by recording the incidence of adverse events.

   1. Record clinical adverse events and clinically significant laboratory abnormalities.
   2. Evaluate overall incidence of adverse events for the study as a whole.
   3. Monitor the incidence of serious adverse events.
2. The primary efficacy objective of this study will be determined by measuring the percentage of subjects who have >= 10% oxidase positive granulocytes by dihydrorhodamine (DHR) flow cytometry at month 6 and 12 after transplant.

Secondary Endpoints:

1. Assess immunological reconstitution:

   Restoration of neutrophil oxidase function (> 10%) as measured by DHR flow cytometry (clinical), and/or cytochrome C (O2 production, research), at 24 months. The % DHR + neutrophils will be measured at week 4, 5, 6, 7, 8, 10, 12 and month 6, 9, 12, 18 and 24.
2. Assess hematopoietic stem cell (HSC) transduction and engraftment:

   1. Determine the percentage of transduced CD34+ hematopoietic cells infused.
   2. Measure the average vector copy number (VCN) in mature blood cells (at week 4, 6, 7, 8, 10, 12 and month 6, 9, 12, 18 and 24) by quantitative polymerase chain reaction (qPCR) or droplet digital polymerase chain reaction (ddPCR).
3. Assess health by:

   1. The nutritional status (height, weight, serum albumin) at 24 months
   2. Growth and development of pediatric subjects at 24 months
   3. Frequency of severe infections or other health issues, including inflammatory complications (requiring intravenous [IV] antibiotics and/or hospitalization for treatment)
   4. Measurement of inflammatory markers at 1, 2, 3, 6, 9, 12, 18, and 24 months, compared to baseline
   5. Colitis assessment based on CDAI (Crohn s Disease Activity Index) and fecal calprotectin at 6, 12, and 24 months, compared to baseline
   6. Quality of Life (QOL) questionnaire (baseline, 6, 12 and 24 months)

Exploratory Endpoints:

1. Evaluation of the human microbiome during XCGD gene therapy
2. Evaluation of inflammatory cytokines and antibody development to Gp91, etc

ELIGIBILITY:
-INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Must have confirmed molecular diagnosis of X-linked CGD confirmed by deoxyribonucleic acid (DNA) sequencing and supported by laboratory evidence for absent or reduction >90% of the biochemical activity of the NADPH-oxidase.
* At least 1 prior ongoing or refractory severe infection and/or inflammatory complications requiring hospitalization despite conventional therapy.
* No 10/10 HLA-matched donor available after initial search of National Marrow Donor Program (NMDP) registries within the last year.
* Must weigh at least 15 kg.
* Male or female, and must be at least 3 years of age but no older than 60.
* Parent/guardian must be willing to sign and date informed consent form for child and where appropriate, child may sign assent.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Ability to take oral medication and be willing to adhere to the prophylactic regimen.
* Apheresis of patients for the hematopoietic stem cells collected as a part of this protocol will be performed according to the Standard of Care apheresis practices established in the NIH CC Department of Transfusion Medicine for such procedures.
* For apheresis, pediatric patients:

  --Must weigh at least 15 kg body weight;

  --Preserved renal function (creatinine <=2.5 mg/dL; <=3+ proteinuria); preserved hepatic function (bilirubin <=2.0 mg/dl);
* Must be negative for co-infection with human immunodeficiency virus (HIV) or hepatitis B virus (HBsAg positive) or hepatitis C virus (HCV ribonucleic acid (RNA) positive), adenovirus, parvovirus B 19 or toxoplasmosis or mycobacterial infection (prior or current).
* For females of reproductive potential, must agree to use of 2 highly effective contraception throughout study participation and for at least 3 months after the study.
* For females:

  * Condoms, male or female, with or without a spermicide;
  * Diaphragm or cervical cap with spermicide;
  * Intrauterine device;
  * Contraceptive pills or patch, Norplant, Depo-Provera, or other FDA- approved contraceptive method;
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner.
* Agreement to adhere to Lifestyle Considerations throughout study duration.
* Ability of subject (Patient/Legal Guardian) to understand and the willingness to sign a written informed consent document.
* For the Natural History Protocol (05-I-0213): All patients must be willing to allow storage of blood samples for future studies.
* Must provide a durable power of attorney (DPA) for health care decisions to an appropriate adult relative or guardian in accordance to NIH-200 "NIH Advance Directive for Health Care and Medical Research Participation."

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Patient/Parent/Guardian unable or unwilling to comply with the protocol requirements.
* Contraindication for leukapheresis (anemia Hb <8 g/dl, cardiovascular instability, severe coagulopathy).
* Patients who are unable to lie prone during the bone marrow harvesting procedure (in the case of bone marrow harvest, contraindication to general anesthesia).
* Have a 10/10 HLA identical (A,B,C,DR,DQ) family or unrelated adult donor unless there is deemed to be an unacceptable risk associated with an allogeneic procedure.
* Tested positive (definitive) for the presence of multiple types (2 or more) of anti-platelet antibodies.
* Altered organ function as outlined below observed within 8 weeks of entering this trial.

  a. Hematologic

  i. Anemia (hemoglobin < 8 g/dl).

ii. Neutropenia (absolute granulocyte count <1,000/mm3 ).

iii. Thrombocytopenia (platelet count < 150,000/mm3).

iv. Prothrombin Time (PT) INR or Partial thromboplastin time (PTT) > 2 X the upper limits of normal (ULN) (patients with a correctable deficiency controlled on medication will not be excluded).

v. Cytogenetic abnormalities known to be associated with hematopoietic defect on peripheral blood or bone marrow.

b. Infectious

i. Evidence of infection with HIV-1 and -2, Hepatitis B, Hepatitis C, adenovirus, parvovirus B 19 or toxoplasmosis within 8 weeks prior to mobilization/apheresis or bone marrow harvest. Cytomegalovirus (CMV) infection is allowable as long as the infection is under control.

ii. History of infection with mycobacteria or Bacille Calmette-Guerin (BCG) vaccination.

c. Pulmonary

i. Resting O2 saturation by pulse oximetry < 90% on room air.

d. Cardiac

i. Abnormal electrocardiogram (ECG) indicating cardiac pathology.

ii. Uncorrected congenital cardiac malformation with clinical symptomatology.

iii. Active cardiac disease, including clinical evidence of congestive heart failure, cyanosis, hypotension.

iv. Poor cardiac function as evidenced by LV ejection fraction <40% on echocardiogram.

e. Neurological

i. Significant neurologic abnormality by examination.

ii. Uncontrolled seizure disorder.

f. Renal

i. Renal insufficiency: serum creatinine >=2.5 mg/dl, or >=3+ proteinuria.

* Chemistry Lab abnormalities: Serum sodium >= 156 mmol/L or <= 129 mmol/L, potassium >= 6.1 mmol/L or <= 2.9 mmol/L, calcium >= 3.2 mmol/L or < 1.74 mmol/L , magnesium >= 1.24 mmol/L or < 0.39 mmol/L, phosphate >= 5.1 mmol/L or < 1.9 mmol/L.
* Serum transaminases > 5X the upper limit of normal (ULN).

Serum bilirubin > 2X the upper limit of normal (ULN).

Serum glucose > 1.5X the upper limit of normal (ULN).

* General

  * Expected survival < 6 months.
  * Major congenital anomaly.
  * Known allergic reactions to components of busulfan or dimethyl sulfoxide (DMSO) or contraindication for administration of conditioning medication.
  * Evidence of active malignant disease.
* Treatment with another investigational drug or other intervention within 6 months.
* Unable to undergo apheresis as per the NIH CC Department of Transfusion Medicine Standard of Care apheresis procedures.

  1. Patients who are hemodynamically unstable (systolic or diastolic blood pressure fall of 20 mm Hg from the stable patient's baseline measurement) or requiring mechanical respiratory assistance are excluded.

History of vasculitis.

* Administration of gamma-interferon within 30 days before the infusion of transduced, autologous CD34+ cells.
* Any other condition that, in the opinion of the Investigator, may compromise the safety or compliance of the patient or would preclude the patient from successful study completion.

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Safety | Throughout the study
  1) The primary safety objective of this procedure will be assessed by recording the incidence of adverse events. a) Record clinical adverse events and clinically significant laboratory abnormalities. b) Evaluate overall incidence of adverse events for the study as a whole. c) Monitor the incidence of serious adverse events.
Efficacy | 6 months and 1 year
  The primary efficacy objective of this study will be determined by measuring the percentage of subjects who have >= 10% oxidase positive granulocytes by DHR flow cytometry at month 6 and 12 after transplant.

SECONDARY OUTCOMES:
Assess immunological reconstitution | Week 4, 5, 6, 7, 8, 10, 12 and months 6, 9, 12, 18 and 24 months.
  Restoration of neutrophil oxidase function (> 10%) as measured by DHR flow cytometry (clinical), and/or cytochrome C (O2 production, research), at 24 months. The % DHR + neutrophils will be measured at week 4, 5, 6, 7, 8, 10, 12 and months 6, 9, 12, 18 and 24 months.
Assess HSC transduction and engraftment | Week 4, 6, 7, 8, 10, 12 and month 6, 9, 12, 18 and 24)
  a) Determine the percentage of transduced CD34+ hematopoietic cells infused. b) Measure the average vector copy number (VCN) in mature blood cells (at week 4, 6, 7, 8, 10, 12 and month 6, 9, 12, 18 and 24) by qPCR or ddPCR.
Assess health by | 1, 2, 3, 6, 9, 12, 18, and 24 months, compared to baseline
  a) The nutritional status (height, weight, serum albumin) at 24 months b) Growth and development of pediatric subjects at 24 months c) Frequency of severe infections or other health issues, including inflammatory complications (requiring IV antibiotics and/or hospitalization for treatment) d) Measurement of inflammatory markers at 1, 2, 3, 6, 9, 12, 18, and 24 months, compared to baseline e) Colitis assessment based on CDAI (Crohn s Disease Activity Index) and fecal calprotectin at 6, 12, and 24 months, compared to baseline f) Quality of life questionnaire (baseline, 6, 12 and 24 months).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Kang, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000186-I.html